CLINICAL TRIAL: NCT03206879
Title: Fecal ESBL Resurgence During Antibiotic Treatment
Status: Terminated | Type: Observational
Why Stopped: Several sites did not manage to recruit patients.
Sponsor: University Hospital, Akershus (Other)
Collaborators: Sorlandet Hospital HF (Other Government); Helse Stavanger HF (Other Government); Sykehuset Telemark (Other Government); Oslo University Hospital (Other); Sykehuset Ostfold (Other)
Responsible Party: Principal Investigator, Silje Bakken Jørgensen, Head of section, infection control officer, University Hospital, Akershus
Other Study IDs: 16-086
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Antibiotic Drug Resistance
Keywords: ESBL; Enterobacteriaceae; multidrug-resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial fecal isolates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Norwegian hospitals are struggling to control spread of extended-spectrum beta-lactamase producing Enterobacteriaceae (ESBL-E) in health care settings. Strict screening and isolation criteria are enforced in hospital, and patients previously infected by ESBL-E are regarded as possible ESBL-E carriers indefinitely. This observational multi-centre cross-sectional study aims to estimate the duration of fecal ESBL-E carriage and to assess the risk of ESBL-E resurgence during hospital stay for patients previously infected by ESBL-E. Through better knowledge of these risk factors, infection control procedures may be better tailored to rhe individual patient.

ELIGIBILITY:
Inclusion Criteria:

Patients with previous infection or colonization with ESBL-E admitted to one of the participating wards. -

Exclusion Criteria:

* Not able to give informed consent.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, hospitalized patients previously infected by ESBL-E.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
fecal carriage of ESBL-E | Baseline

SECONDARY OUTCOMES:
fecal ESBL-E carriage developed during admission | Baseline (admission)

CONTACTS AND LOCATIONS:
Overall Officials: Silje B Jørgensen, MD, Principal Investigator — Akershus univversitetssykehus HF

IPD SHARING:
Plan to Share IPD: No